CLINICAL TRIAL: NCT03937479
Title: A Phase II, Randomized, Double-Blind, Placebo Controlled Dose Ranging Study to Assess the Effect of RPL554 Added on to Tiotropium in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Study Investigating the Effect of 4 Doses of RPL554 Given in Addition to Tiotropium to Patients With COPD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Verona Pharma plc (Industry)
Collaborators: Iqvia Pty Ltd (Industry); LGC Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RPL554-CO-205
Record Dates: First submitted 2019-05-01; First posted 2019-05-03 (Actual); Results first posted 2020-10-28 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-10

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — ensifentrine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- RPL554 0.375 mg twice daily (Experimental): RPL554 0.375 mg twice daily
  Interventions: Drug: Ensifentrine (formerly RPL554) 0.375 mg twice daily plus placebo, in addition to tiotropium
- RPL554 0.75 mg twice daily (Experimental): RPL554 0.75 mg twice daily
  Interventions: Drug: Ensifentrine (formerly RPL554) 0.75 mg twice daily plus placebo, in addition to tiotropium
- RPL554 1.5 mg twice daily (Experimental): RPL554 1.5 mg twice daily
  Interventions: Drug: Ensifentrine (formerly RPL554) 1.5 mg twice daily plus placebo, in addition to tiotropium
- RPL554 3.0 mg twice daily (Experimental): RPL554 3.0 mg twice daily
  Interventions: Drug: Ensifentrine (formerly RPL554) 3.0 mg twice daily plus placebo, in addition to tiotropium
- Placebo twice daily (Placebo Comparator): Placebo twice daily
  Interventions: Drug: Ensifentrine (formerly RPL554) placebo twice daily, in addition to tiotropium

INTERVENTIONS:
Drug: Ensifentrine (formerly RPL554) 0.375 mg twice daily plus placebo, in addition to tiotropium — Patients will be randomized to receive one of the following treatment arms plus tiotropiuim:
  ● RPL554 0.375 mg twice daily The approximate planned duration for each completed patient will be 14 days of run-in and 28 days of treatment with study medication.
  Arms: RPL554 0.375 mg twice daily
Drug: Ensifentrine (formerly RPL554) 0.75 mg twice daily plus placebo, in addition to tiotropium — Patients will be randomized to receive one of the following treatment arms plus tiotropiuim:
  ● RPL554 0.75 mg twice daily The approximate planned duration for each completed patient will be 14 days of run-in and 28 days of treatment with study medication.
  Arms: RPL554 0.75 mg twice daily
Drug: Ensifentrine (formerly RPL554) 1.5 mg twice daily plus placebo, in addition to tiotropium — Patients will be randomized to receive one of the following treatment arms plus tiotropiuim:
  ● RPL554 1.5 mg twice daily The approximate planned duration for each completed patient will be 14 days of run-in and 28 days of treatment with study medication.
  Arms: RPL554 1.5 mg twice daily
Drug: Ensifentrine (formerly RPL554) 3.0 mg twice daily plus placebo, in addition to tiotropium — Patients will be randomized to receive one of the following treatment arms plus tiotropiuim:
  ● RPL554 3.0 mg twice daily The approximate planned duration for each completed patient will be 14 days of run-in and 28 days of treatment with study medication.
  Arms: RPL554 3.0 mg twice daily
Drug: Ensifentrine (formerly RPL554) placebo twice daily, in addition to tiotropium — Patients will be randomized to receive one of the following treatment arms plus tiotropiuim:
  ● Placebo twice daily The approximate planned duration for each completed patient will be 14 days of run-in and 28 days of treatment with study medication.
  Arms: Placebo twice daily

SUMMARY:
The purpose of this study is to investigate the dose response of RPL554 in patients with moderate to severe CHRONIC OBSTRUCTIVE PULMONARY DISEASE that are still symptomatic despite treatment with a stable background of tiotropium over 4 weeks of treatment. This study is intended to support optimal dose selection for a Phase III program evaluating RPL554 as an add-on treatment to standard of care therapy.

DETAILED DESCRIPTION:
This is a Phase IIb, randomized, double-blind, placebo controlled, multiple dose, parallel group study to investigate the effects of 4 weeks of treatment with nebulized RPL554 (at different dose levels) compared to placebo in patients with moderate to severe CHRONIC OBSTRUCTIVE PULMONARY DISEASE on a stable background therapy of open-label tiotropium. The study comprises seven visits: Pre-screening (Visit 0), Screening (Visit 1) and then a Treatment Period consisting of Randomization (Visit 2), and weekly visits for 4 weeks (Visit 3 to Visit 6).

ELIGIBILITY:
Inclusion Criteria:

* Sign an informed consent document indicating they understand the purpose of and procedures required for the study and are willing to participate in the study.
* Male or female aged between 40 and 80 years inclusive, at the time of informed consent.
* Must agree to meet the following from the first dose up to 1 month after the last dose of study medication:

  * If male:

    * Not donate sperm
    * Either: be sexually abstinent in accordance with a patient's usual and preferred lifestyle (but agree to abide by the contraception requirements below should their circumstances change)
    * Or: use a condom with all sexual partners. If the partner is of childbearing potential the condom must be used with spermicide and a second reliable form of contraception must also be used (e.g., diaphragm/cap with spermicide, established hormonal contraception, intra-uterine device)
  * If female:

    * be of non-childbearing potential or use a highly effective form of contraception
* Have a 12-lead ECG recording at Screening showing the following (and no changes in the pre-dose value at the first treatment deemed clinically significant by the Investigator):

  * Heart rate between 45 and 90 beats per minute
  * QT interval corrected for heart rate using Fridericia's formula (QTcF) ≤450 msec for males, and ≤ 470 msec for females
  * QRS interval ≤ 120 msec
  * No clinically significant abnormality including morphology (e.g., left bundle branch block, atrio-ventricular nodal dysfunction, ST segment abnormalities consistent with ischemia)
* Capable of complying with study restrictions and procedures, including ability to use the nebulizer correctly.
* Body mass index (BMI) between 18 and 35 kg/m2 (inclusive) with a minimum weight of 45 kg.
* COPD diagnosis: Patients with a diagnosis of COPD as defined by the American Thoracic Society (ATS)/European Respiratory Society (ERS) guidelines (Celli and MacNee, 2004) with symptoms compatible with COPD for at least 1 year prior to Screening.
* Ability to perform acceptable and reproducible spirometry.
* Post-bronchodilator (four puffs of albuterol) spirometry at Screening demonstrating the following:

  * FEV1/ FVC ratio of ≤0.70
  * FEV1 ≥30% and ≤70% of predicted normal* *National Health and Nutrition Examination Survey (NHANES) III (Hankinson et al, 1999) will be used as the reference for normal predicted values.
* Clinically stable COPD in the 4 weeks prior to Screening (Visit 1) and during the period between Visits 1 and 2.
* A score of ≥2 on the modified Medical Research Council (mMRC) dyspnea scale at Screening.
* A chest X-ray (posterior-anterior) at Screening, or in the 12 months prior to Screening showing no clinically significant abnormalities unrelated to COPD.
* Meet the concomitant medication restrictions and be expected to do so for the rest of the study.
* Current and former smokers with smoking history of ≥10 pack years.
* Capable of withdrawing from long acting bronchodilators (other than tiotropium) for the duration of the study, and short acting bronchodilators for 6 hours prior to dosing.

Exclusion Criteria:

* A history of life-threatening COPD including Intensive Care Unit admission and/or requiring intubation.
* COPD exacerbation requiring oral or parenteral steroids, or lower respiratory tract infection requiring antibiotics, within 3 months of Screening or prior to the first treatment.
* A history of one or more hospitalizations for COPD or pneumonia within 6 months of Screening or prior to the first treatment.
* Intolerance or hypersensitivity to albuterol, tiotropium or other muscarinic receptor antagonists.
* Other respiratory disorders: Patients with a current diagnosis of asthma, active tuberculosis, lung cancer, bronchiectasis, sarcoidosis, lung fibrosis, interstitial lung diseases, uncontrolled or unstable sleep apnea, known alpha-1 antitrypsin deficiency, core pulmonale, clinically significant pulmonary hypertension or other active pulmonary diseases.
* Previous lung resection or lung reduction surgery.
* Pulmonary rehabilitation, unless such treatment has been stable from 4 weeks prior to Screening and remains stable during the study.
* Oral therapies for COPD (e.g. oral steroids, theophylline, and roflumilast) or antibiotics within 3 months prior to Screening, or ICS therapy within 4 weeks prior to Screening
* Prior exposure to RPL554.
* History of, or reason to believe a patient has, drug or alcohol abuse within the past 5 years.
* Received an experimental drug within 30 days or five half-lives, whichever is longer.
* Women who are pregnant or breast-feeding.
* Patients with uncontrolled disease including, but not limited to, endocrine, active hyperthyroidism, neurological, hepatic, gastrointestinal, renal, hematological, urological, immunological, psychiatric, or ophthalmic diseases that the Investigator believes are clinically significant. This includes any hepatic disease or moderate to severe renal impairment.
* Documented clinically significant cardiovascular disease such as: any history of arrhythmias, angina, recent (<1 year) or suspected myocardial infarction, congestive heart failure, unstable or uncontrolled hypertension, or diagnosis of hypertension within 3 months prior to Screening.
* Use of non-selective oral β-blockers.
* Major surgery (requiring general anesthesia) within 6 weeks prior to Screening, lack of full recovery from surgery at Screening, or planned surgery through the end of the study.
* Required use of oxygen therapy, even on an occasional basis.
* History of malignancy of any organ system within 5 years, with the exception of localized skin cancers (basal or squamous cell).
* Clinically significant abnormal values for laboratory safety tests (hematology, blood chemistry, viral serology or urinalysis) at Screening, as determined by the Investigator. In particular, alanine aminotransferase or aspartate aminotransferase cannot be more than twice the upper limit of normal.
* Patients with conditions which are sensitive to antimuscarinic effects such as narrow angle glaucoma, urinary retention, prostatic hypertrophy, or bladder neck obstruction.
* Current marijuana use (all forms).
* A disclosed history or one known to the Investigator, of significant non-compliance in previous investigational studies or with prescribed medications.
* Any other reason that the Investigator considers makes the patient unsuitable to participate.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 416 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2019-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Ferguson, Principal Investigator — Pulmonary Research Institute of Southeast Michigan
Locations (50):
- United States (50):
  - Pinnacle Research Group, LLC, Anniston, Alabama
  - California Research Medical Group, Inc, Fullerton, California
  - Southern California Institute For Respiratory Diseases, Inc., Los Angeles, California
  - Innovative Clinical Research, Lafayette, Colorado
  - Meris Clinical Research, Brandon, Florida
  - Clinical Research of West Florida, Clearwater, Florida
  - Pulmonary Disease Specialists, PA d/b/a PDS Research, Kissimmee, Florida
  - Medical Research of Central Florida, LLC, Leesburg, Florida
  - Clinical Trials of Florida, LLC, Miami, Florida
  - Peninsula Research, Ormond Beach, LLC, Ormond Beach, Florida
  - Medsol Clinical Research Center, Inc, Port Charlotte, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Pasadena Center for Medical Research, LLC, St. Petersburg, Florida
  - Florida Pulmonary Research Institute, LLC, Winter Park, Florida
  - Columbus Regional Research Institute, Columbus, Georgia
  - VitaLink Research - Hamilton Mill, Dacula, Georgia
  - VitaLink Research - Duluth, Duluth, Georgia
  - Gwinnett Biomedical Research, Lawrenceville, Georgia
  - IACT Health, Rincon, Georgia
  - Vitalink, Winder, Georgia
  - Genesis Clinical Research and Consulting, LLC, Fall River, Massachusetts
  - Pulmonary Research Institute of Southeast Michigan, Farmington Hills, Michigan
  - Cities Research Center, Fridley, Minnesota
  - American Health Research, Charlotte, North Carolina
  - Clinical Research of Gastonia, Gastonia, North Carolina
  - Research Carolina of Huntersville, Huntersville, North Carolina
  - Clinical Research of Lake Norman, Mooresville, North Carolina
  - New Horizons Clinical Research, Cincinnati, Ohio
  - Aventiv Research, Inc, Columbus, Ohio
  - Aventiv Research, Inc, Dublin, Ohio
  - Crisor, LLC, Medford, Oregon
  - Vitalink Research - Anderson, Anderson, South Carolina
  - Lowcountry Lung and Critical Care, PA, Charleston, South Carolina
  - VitaLink-Columbia, Columbia, South Carolina
  - VitaLink Research - Easley, Easley, South Carolina
  - Piedmont Research Partners, LLC, Fort Mill, South Carolina
  - VitaLink Research-Gaffney, Gaffney, South Carolina
  - VitaLink Research-Greenville, Greenville, South Carolina
  - VitaLink Research-UPSTATE, Greenville, South Carolina
  - Clinical Research of Charleston, Mt. Pleasant, South Carolina
  - Clinical Research of Rock Hill, Rock Hill, South Carolina
  - Vitalink Research-Seneca, Seneca, South Carolina
  - Fusion Clinical Research of Spartanburg, LLC, Spartanburg, South Carolina
  - Spartanburg Medical Research, Spartanburg, South Carolina
  - Vitalink Research-Spartanburg, Spartanburg, South Carolina
  - VitaLink Research - Union, Union, South Carolina
  - New Phase Research & Development, Knoxville, Tennessee
  - FMC Science, LLC, Lampasas, Texas
  - DCOL Center for Clinical Research, Longview, Texas
  - Metroplex Pulmonary and Sleep Center, McKinney, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 49 study centers in the United States of America between 01 May 2019 and 15 November 2019. Overall, 416 adult patients with moderate to severe chronic obstructive pulmonary disease (COPD) on a stable background therapy of open-label tiotropium were randomized and 413 patients received double-blind study treatment.
Pre-assignment Details: Following Screening on Visit 1, eligible patients entered a 14-day run-in period, where they received tiotropium once daily. At Visit 2, patients were re-assessed for eligibility according to randomization criteria. Patients were randomized equally across 5 double-blind treatment groups (4 doses of RPL554 or placebo).
Groups:
- RPL554 0.375 mg: Patients were administered 0.375 milligram (mg) RPL554 by jet nebulizer twice daily (morning and evening) for 4 weeks. Open-label tiotropium was administered once daily in the morning.
- RPL554 0.75 mg: Patients were administered 0.75 mg RPL554 by jet nebulizer twice daily (morning and evening) for 4 weeks. Open-label tiotropium was administered once daily in the morning.
- RPL554 1.5 mg: Patients were administered 1.5 mg RPL554 by jet nebulizer twice daily (morning and evening) for 4 weeks. Open-label tiotropium was administered once daily in the morning.
- RPL554 3.0 mg: Patients were administered 3.0 mg RPL554 by jet nebulizer twice daily (morning and evening) for 4 weeks. Open-label tiotropium was administered once daily in the morning.
- Placebo: Patients were administered placebo (matching with RPL554) by jet nebulizer twice daily (morning and evening) for 4 weeks. Open-label tiotropium was administered once daily in the morning.
Period: Overall Study
Arm/Group | RPL554 0.375 mg | RPL554 0.75 mg | RPL554 1.5 mg | RPL554 3.0 mg | Placebo
Started | 83 | 85 | 82 | 82 | 84
Received Treatment | 83 | 83 | 81 | 82 | 84
Completed | 73 | 70 | 75 | 76 | 79
Not Completed | 10 | 15 | 7 | 6 | 5
Not completed — Adverse Event | 2 | 3 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 3 | 5 | 2 | 2 | 1
Not completed — Protocol Violation | 5 | 6 | 4 | 3 | 2
Not completed — Lost to Follow-up | 0 | 1 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All Patients Randomized Set included all patients who provided informed consent and who were randomized to study treatment.
Groups:
- RPL554 0.375 mg: Patients were administered 0.375 mg RPL554 by jet nebulizer twice daily (morning and evening) for 4 weeks. Open-label tiotropium was administered once daily in the morning.
- Total: Total of all reporting groups
Arm/Group | RPL554 0.375 mg | RPL554 0.75 mg | RPL554 1.5 mg | RPL554 3.0 mg | Placebo | Total
Number analyzed (Participants) | 83 | 85 | 82 | 82 | 84 | 416
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 44 | 40 | 45 | 41 | 47 | 217
  >=65 years | 39 | 45 | 37 | 41 | 37 | 199
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.2 (7.86) | 65.5 (8.33) | 63.8 (7.67) | 64.5 (7.92) | 63.6 (8.41) | 64.3 (8.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 48 | 51 | 45 | 44 | 239
  Male | 32 | 37 | 31 | 37 | 40 | 177
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 2 | 3 | 8
  Not Hispanic or Latino | 82 | 84 | 81 | 80 | 81 | 408
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 10 | 7 | 9 | 6 | 9 | 41
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  White | 73 | 78 | 73 | 76 | 75 | 375
  Other | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Least Square (LS) Mean Change From Baseline Forced Expiratory Volume in 1 Second (FEV1) to Peak FEV1 at Week 4
Description: Forced spirometry maneuvers including the FEV1 were used to assess pulmonary function. Baseline FEV1 was defined as the value of FEV1 assessed 30 minutes before first administration and peak FEV1 was defined as the maximum value in the 3 hours after dosing. Spirometry assessments were performed in accordance with American Thoracic Society (ATS)/European Respiratory Society (ERS) guidelines.
Time Frame: Baseline and Week 4
Population: The Full Analysis Set (FAS) included all randomized patients with sufficient data collected after intake of study treatment to compute any of the FEV1 parameters on at least 1 occasion. Only patients with valid values at baseline and Week 4 are included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | RPL554 0.375 mg | RPL554 0.75 mg | RPL554 1.5 mg | RPL554 3.0 mg | Placebo
Number analyzed (Participants) | 73 | 70 | 75 | 76 | 79
liters | 0.1963 (0.02639) | 0.2100 (0.02676) | 0.2260 (0.02647) | 0.2431 (0.02631) | 0.1188 (0.02589)
Statistical Analysis 1: Comparison: RPL554 3.0 mg vs Placebo; Comparison was done using a closed testing procedure; testing began at the highest dose of RPL554 compared with placebo. If found statistically significant then the next highest dose was compared with placebo. This continued until a result was found to be non-significant or all RPL554 doses were compared with placebo; Test type: Superiority; p = 0.0008, MMRM — The mixed model for repeated measures (MMRM) model was used to model the change from baseline FEV1 to peak FEV1 using treatment, visit and treatment by visit interaction as fixed effect, patient as random effect and baseline FEV1 as the covariate; LS mean difference = 0.1242, 95% CI 2-sided [0.0517 to 0.1968], Standard Error of Mean 0.03691 — Estimates refer to the Week 4 from treatment by visit interaction
Statistical Analysis 2: Comparison: RPL554 1.5 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0040, MMRM — The MMRM model was used to model the change from baseline FEV1 to peak FEV1 using treatment, visit and treatment by visit interaction as fixed effect, patient as random effect and baseline FEV1 as the covariate; LS mean difference = 0.1072, 95% CI 2-sided [0.0344 to 0.1800], Standard Error of Mean 0.03703 — Estimates refer to the Week 4 from treatment by visit interaction
Statistical Analysis 3: Comparison: RPL554 0.75 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0148, MMRM — [p-value comment as in outcome 1, analysis 2]; LS mean difference = 0.0912, 95% CI 2-sided [0.0180 to 0.1643], Standard Error of Mean 0.03723 — Estimates refer to the Week 4 from treatment by visit interaction
Statistical Analysis 4: Comparison: RPL554 0.375 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0368, MMRM — [p-value comment as in outcome 1, analysis 2]; LS mean difference = 0.0775, 95% CI 2-sided [0.0048 to 0.1501], Standard Error of Mean 0.03697 — Estimates refer to the Week 4 from treatment by visit interaction

2. Secondary Outcome: LS Mean Change From Baseline FEV1 to Average Area Under the Curve Over 3 Hours (AUC0-3h) FEV1 on Day 1 and at Weeks 1 to 4
Description: Forced spirometry maneuvers including the FEV1 were used to assess pulmonary function. Baseline FEV1 was defined as the value of FEV1 assessed 30 minutes before first administration and average AUC0-3h FEV1 was defined as area under the curve over 3 hours of the FEV1, divided by 3 hours. Spirometry assessments were performed in accordance with ATS/ERS guidelines.
Time Frame: Baseline (30 minutes before first administration on Day 1); 30 minutes and 1, 2, and 3 hours post-dose on Day 1 and Weeks 1, 2, 3 and 4
Population: The FAS included all randomized patients with sufficient data collected after intake of study treatment to compute any of the FEV1 parameters on at least 1 occasion. Number of patients with valid values at baseline and at the specific visit were analyzed.
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | RPL554 0.375 mg | RPL554 0.75 mg | RPL554 1.5 mg | RPL554 3.0 mg | Placebo
Number analyzed (Participants) | 83 | 83 | 81 | 82 | 84
liters
  Day 1 | 0.1533 (0.01600) | 0.1614 (0.01602) | 0.1810 (0.01620) | 0.2017 (0.01609) | 0.0654 (0.01590)
  Week 1: number analyzed (Participants) | 80 | 78 | 80 | 78 | 82
  Week 1 | 0.1118 (0.02129) | 0.1301 (0.02144) | 0.1308 (0.02143) | 0.1526 (0.02149) | 0.0246 (0.02107)
  Week 2: number analyzed (Participants) | 78 | 74 | 76 | 78 | 80
  Week 2 | 0.1154 (0.02308) | 0.1309 (0.02338) | 0.1433 (0.02334) | 0.1651 (0.02321) | 0.0304 (0.02285)
  Week 3: number analyzed (Participants) | 76 | 71 | 75 | 78 | 78
  Week 3 | 0.1156 (0.02323) | 0.1243 (0.02364) | 0.1444 (0.02343) | 0.1385 (0.02324) | 0.0294 (0.02297)
  Week 4: number analyzed (Participants) | 73 | 70 | 75 | 76 | 79
  Week 4 | 0.1095 (0.02538) | 0.1305 (0.02574) | 0.1394 (0.02544) | 0.1626 (0.02530) | 0.0369 (0.02488)

3. Secondary Outcome: LS Mean Change From Baseline FEV1 to Average Area Under the Curve Over 12 Hours (AUC0-12h) FEV1 on Day 1 and at Week 4
Description: Forced spirometry maneuvers including the FEV1 were used to assess pulmonary function. Baseline FEV1 was defined as the value of FEV1 assessed 30 minutes before first administration and average AUC0-12h FEV1 was defined as area under the curve over 12 hours of the FEV1, divided by 12 hours. Spirometry assessments were performed in accordance with ATS/ERS guidelines.
Time Frame: Baseline (30 minutes before first administration on Day 1); 30 minutes and 1, 2, 3, 4, 6, 8 and 12 hours post-dose on Day 1 and at Week 4
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | RPL554 0.375 mg | RPL554 0.75 mg | RPL554 1.5 mg | RPL554 3.0 mg | Placebo
Number analyzed (Participants) | 83 | 83 | 81 | 82 | 84
liters
  Day 1 | 0.0795 (0.01767) | 0.0909 (0.01770) | 0.1020 (0.01790) | 0.1374 (0.01777) | 0.0282 (0.01756)
  Week 4: number analyzed (Participants) | 74 | 71 | 76 | 78 | 78
  Week 4 | 0.0359 (0.02455) | 0.0630 (0.02486) | 0.0640 (0.02451) | 0.0969 (0.02426) | 0.0096 (0.02413)

4. Secondary Outcome: LS Mean Change From Baseline FEV1 to Peak FEV1 on Day 1 and at Weeks 1 to 3
Description: Forced spirometry maneuvers including the FEV1 were used to assess pulmonary function. Baseline FEV1 was defined as the value of FEV1 assessed 30 minutes before first administration and peak FEV1 was defined as the maximum value in the 3 hours after dosing. Spirometry assessments were performed in accordance with ATS/ERS guidelines.
Time Frame: Baseline (30 minutes before first administration on Day 1); 30 minutes post-dose on Day 1 and Weeks 1, 2 and 3
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | RPL554 0.375 mg | RPL554 0.75 mg | RPL554 1.5 mg | RPL554 3.0 mg | Placebo
Number analyzed (Participants) | 83 | 83 | 81 | 82 | 84
liters
  Day 1 | 0.2353 (0.01926) | 0.2426 (0.01930) | 0.2610 (0.01951) | 0.2852 (0.01938) | 0.1469 (0.01914)
  Week 1: number analyzed (Participants) | 80 | 78 | 80 | 78 | 83
  Week 1 | 0.1860 (0.02305) | 0.2026 (0.02322) | 0.2116 (0.02321) | 0.2353 (0.02326) | 0.1041 (0.02277)
  Week 2: number analyzed (Participants) | 78 | 74 | 76 | 78 | 80
  Week 2 | 0.1963 (0.02453) | 0.2121 (0.02483) | 0.2191 (0.02481) | 0.2421 (0.02466) | 0.1098 (0.02429)
  Week 3: number analyzed (Participants) | 76 | 71 | 75 | 78 | 78
  Week 3 | 0.1987 (0.02503) | 0.2006 (0.02544) | 0.2277 (0.02526) | 0.2197 (0.02505) | 0.1072 (0.02476)

5. Secondary Outcome: LS Mean Change From Baseline FEV1 to Morning Trough FEV1 at Weeks 1 to 4
Description: Forced spirometry maneuvers including the FEV1 were used to assess pulmonary function. Baseline FEV1 was defined as the value of FEV1 assessed 30 minutes before first administration and morning trough FEV1 was defined as the last pre-dose value. Spirometry assessments were performed in accordance with ATS/ERS guidelines.
Time Frame: Baseline (30 minutes before first administration on Day 1) and morning pre-dose on Weeks 1, 2, 3 and 4
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | RPL554 0.375 mg | RPL554 0.75 mg | RPL554 1.5 mg | RPL554 3.0 mg | Placebo
Number analyzed (Participants) | 83 | 83 | 81 | 82 | 84
liters
  Week 1: number analyzed (Participants) | 81 | 80 | 80 | 78 | 82
  Week 1 | -0.0088 (0.02038) | -0.0354 (0.02058) | -0.0451 (0.02056) | -0.0216 (0.02081) | -0.0520 (0.02024)
  Week 2: number analyzed (Participants) | 80 | 75 | 78 | 78 | 81
  Week 2 | -0.0278 (0.02183) | -0.0696 (0.02243) | -0.0070 (0.02212) | 0.0136 (0.02220) | -0.0377 (0.02169)
  Week 3: number analyzed (Participants) | 78 | 72 | 75 | 78 | 80
  Week 3 | -0.0385 (0.02185) | -0.0630 (0.02254) | -0.0413 (0.02222) | -0.0232 (0.02205) | -0.0533 (0.02162)
  Week 4: number analyzed (Participants) | 75 | 71 | 75 | 76 | 79
  Week 4 | -0.0201 (0.02296) | -0.0348 (0.02356) | -0.0141 (0.02311) | 0.0054 (0.02306) | -0.0218 (0.02256)

6. Secondary Outcome: LS Mean Change From Baseline to the Mean Weekly Evaluating Respiratory Symptoms of COPD (E-RS:COPD) Total Score at Weeks 1 to 4
Description: The E-RS scale consists of 11 questions, with 3 sub-domains of: breathlessness, cough and sputum, and chest symptoms. The E-RS sub-domain score was calculated as the sum from the relevant questions. The E-RS:COPD scale has a scoring range of 0 to 40. Higher scores indicates severe respiratory symptoms. Baseline was the mean over the 7 days prior to first intake of study treatment. Scores were derived weekly as the mean over 7 days prior to the visit, using only days where data was recorded. The E-RS:COPD was measured by daily electronic diary (e-diary).
Time Frame: Baseline and Weeks 1, 2, 3 and 4
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | RPL554 0.375 mg | RPL554 0.75 mg | RPL554 1.5 mg | RPL554 3.0 mg | Placebo
Number analyzed (Participants) | 83 | 83 | 81 | 82 | 84
units on a scale
  Week 1: number analyzed (Participants) | 82 | 82 | 80 | 80 | 82
  Week 1 | -0.978 (0.3375) | -0.669 (0.3375) | -0.617 (0.3403) | -1.142 (0.3405) | -0.319 (0.3397)
  Week 2: number analyzed (Participants) | 78 | 76 | 79 | 75 | 81
  Week 2 | -0.873 (0.3916) | -0.471 (0.3932) | -0.597 (0.3921) | -0.598 (0.3952) | -0.102 (0.3908)
  Week 3: number analyzed (Participants) | 75 | 72 | 74 | 77 | 75
  Week 3 | -0.950 (0.3830) | -0.338 (0.3865) | -1.091 (0.3843) | -1.097 (0.3827) | -0.287 (0.3832)
  Week 4: number analyzed (Participants) | 75 | 69 | 75 | 74 | 77
  Week 4 | -1.690 (0.4337) | -0.593 (0.4412) | -1.226 (0.4346) | -1.071 (0.4357) | -0.228 (0.4320)

7. Secondary Outcome: LS Mean Change From Baseline in the St George's Respiratory Questionnaire - COPD Specific (SGRQ-C) Total Score at Weeks 2 and 4
Description: Patients completed the SGRQ-C consisting of 40 items each weighted from 0 to a possible maximum of 100. Items 1-7 produced the symptoms score, 9-12 the activity score, and items 8, 10, 11, 13 and 14 the impacts score. Each component sub-score was calculated as a percentage of the summed weights of each item out of the sum of the maximum possible weight for that component (range 0-100). The total score was calculated by summing the weights to all positive responses in each component, where a positive item indicated the presence of symptoms, expressed as a percentage (range 0-100). Higher scores indicated a worse outcome. The SGRQ-C was measured at Week 2 and 4 visits.
Time Frame: Baseline, Weeks 2 and 4
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | RPL554 0.375 mg | RPL554 0.75 mg | RPL554 1.5 mg | RPL554 3.0 mg | Placebo
Number analyzed (Participants) | 83 | 83 | 81 | 82 | 84
units on a scale
  Week 2: number analyzed (Participants) | 79 | 72 | 75 | 73 | 75
  Week 2 | -1.808 (1.1960) | -1.132 (1.2583) | -3.465 (1.2311) | -3.618 (1.2491) | -0.249 (1.2277)
  Week 4: number analyzed (Participants) | 75 | 69 | 71 | 73 | 76
  Week 4 | -4.387 (1.3087) | -2.400 (1.3732) | -4.870 (1.3480) | -4.163 (1.3479) | -0.116 (1.3195)

8. Secondary Outcome: LS Mean Transition Dyspnea Index (TDI) Questionnaire Total Score at Weeks 2 and 4
Description: The TDI is a questionnaire that focussed on 3 sub-domains: functional impairment, magnitude of task and magnitude of effort. Sub-domain score was calculated as the sum from the related questions. Total score was calculated as the sum of the sub-domain scores. The TDI measures the change in dyspnea severity from the baseline as measured by the baseline dyspnea index. It was rated by 7 grades ranging from -3 (major deterioration) to +3 (major improvement). Higher scores indicate better outcome.
Time Frame: Weeks 2 and 4
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | RPL554 0.375 mg | RPL554 0.75 mg | RPL554 1.5 mg | RPL554 3.0 mg | Placebo
Number analyzed (Participants) | 83 | 83 | 81 | 82 | 84
units on a scale
  Week 2: number analyzed (Participants) | 81 | 77 | 79 | 78 | 80
  Week 2 | 1.682 (0.3183) | 1.285 (0.3263) | 1.582 (0.3229) | 1.589 (0.3255) | 1.421 (0.3202)
  Week 4: number analyzed (Participants) | 77 | 74 | 75 | 78 | 80
  Week 4 | 2.089 (0.3423) | 1.484 (0.3496) | 2.055 (0.3475) | 2.063 (0.3437) | 1.766 (0.3381)

9. Secondary Outcome: LS Mean Patient Global Assessment of Change (PGAC) Questionnaire Total Score at Weeks 2 and 4
Description: The PGAC is a single question assessment to determine whether patients noticed a change in their breathing since the start of the study. Patients were asked to respond to a PGAC question asking, "Compared with prior to the study start, how do you feel your breathing is?" on a scale of '1=much worse' to '5=much better', with '3=no change'. Higher scores indicate better outcome.
Time Frame: Weeks 2 and 4
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | RPL554 0.375 mg | RPL554 0.75 mg | RPL554 1.5 mg | RPL554 3.0 mg | Placebo
Number analyzed (Participants) | 83 | 83 | 81 | 82 | 84
units on a scale
  Week 2: number analyzed (Participants) | 80 | 75 | 79 | 76 | 78
  Week 2 | 3.512 (0.0867) | 3.522 (0.0895) | 3.456 (0.0876) | 3.523 (0.0889) | 3.427 (0.0876)
  Week 4: number analyzed (Participants) | 76 | 73 | 75 | 78 | 80
  Week 4 | 3.553 (0.0922) | 3.543 (0.0944) | 3.536 (0.0932) | 3.577 (0.0922) | 3.506 (0.0909)

10. Secondary Outcome: LS Mean Change From Baseline to the Mean Weekly Values Over Weeks 1 to 4 in Number of Puffs of Rescue Medication
Description: Use of rescue medication (albuterol) per visit was calculated as the LS mean use daily over total number of days between previous visit (inclusive) and the following visit. Baseline use was the mean over the last 7 days of the run-in phase (calculated as the sum of puffs taken, divided by number of days data has been recorded).
Time Frame: Baseline and Weeks 1, 2, 3 and 4
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: number of rescue medication puffs
Arm/Group | RPL554 0.375 mg | RPL554 0.75 mg | RPL554 1.5 mg | RPL554 3.0 mg | Placebo
Number analyzed (Participants) | 83 | 83 | 81 | 82 | 84
number of rescue medication puffs
  Week 1: number analyzed (Participants) | 81 | 77 | 79 | 76 | 81
  Week 1 | -0.510 (0.1384) | -0.580 (0.1407) | -0.539 (0.1395) | -0.629 (0.1412) | -0.556 (0.1386)
  Week 2: number analyzed (Participants) | 77 | 75 | 77 | 73 | 80
  Week 2 | -0.325 (0.1822) | -0.360 (0.1847) | -0.388 (0.1828) | -0.379 (0.1850) | -0.544 (0.1812)
  Week 3: number analyzed (Participants) | 75 | 69 | 73 | 74 | 74
  Week 3 | -0.302 (0.1726) | -0.139 (0.1765) | -0.647 (0.1736) | -0.558 (0.1742) | -0.504 (0.1724)
  Week 4: number analyzed (Participants) | 74 | 68 | 72 | 71 | 76
  Week 4 | -0.412 (0.1753) | -0.510 (0.1799) | -0.784 (0.1766) | -0.506 (0.1777) | -0.671 (0.1741)

11. Secondary Outcome: LS Mean Change From Baseline Forced Vital Capacity (FVC) to Peak FVC on Day 1 and at Weeks 1 to 4
Description: Forced spirometry maneuvers including the FVC were used to assess pulmonary function. Baseline FVC was defined as the value of FVC assessed 30 minutes before first administration and peak FVC was defined as the maximum value in the 3 hours after dosing. Spirometry assessments were performed in accordance with ATS/ERS guidelines.
Time Frame: Baseline (30 minutes before first administration on Day 1); 30 minutes post-dose on Day 1 and Weeks 1, 2, 3 and 4
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | RPL554 0.375 mg | RPL554 0.75 mg | RPL554 1.5 mg | RPL554 3.0 mg | Placebo
Number analyzed (Participants) | 83 | 83 | 81 | 82 | 84
liters
  Day 1 | 0.3463 (0.02857) | 0.3775 (0.02858) | 0.3852 (0.02892) | 0.4035 (0.02874) | 0.2241 (0.02840)
  Week 1: number analyzed (Participants) | 80 | 78 | 80 | 78 | 83
  Week 1 | 0.2839 (0.03281) | 0.3199 (0.03302) | 0.3065 (0.03302) | 0.3545 (0.03311) | 0.1717 (0.03242)
  Week 2: number analyzed (Participants) | 78 | 74 | 76 | 78 | 80
  Week 2 | 0.2597 (0.03401) | 0.3282 (0.03446) | 0.3070 (0.03440) | 0.3343 (0.03417) | 0.1524 (0.03368)
  Week 3: number analyzed (Participants) | 76 | 71 | 75 | 78 | 78
  Week 3 | 0.2744 (0.03512) | 0.3177 (0.03570) | 0.3176 (0.03544) | 0.3008 (0.03513) | 0.1626 (0.03475)
  Week 4: number analyzed (Participants) | 73 | 70 | 75 | 76 | 79
  Week 4 | 0.2706 (0.03724) | 0.3198 (0.03775) | 0.2951 (0.03729) | 0.3414 (0.03707) | 0.1736 (0.03647)

12. Secondary Outcome: LS Mean Change From Baseline FVC to Average AUC0-3h FVC on Day 1 and at Weeks 1 to 4
Description: Forced spirometry maneuvers including the FVC were used to assess pulmonary function. Baseline FVC was defined as the value of FVC assessed 30 minutes before first administration and average AUC0-3h FVC was defined as area under the curve over 3 hours of the FVC, divided by 3 hours. Spirometry assessments were performed in accordance with ATS/ERS guidelines.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | RPL554 0.375 mg | RPL554 0.75 mg | RPL554 1.5 mg | RPL554 3.0 mg | Placebo
Number analyzed (Participants) | 83 | 83 | 81 | 82 | 84
liters
  Day 1 | 0.2165 (0.02390) | 0.2397 (0.02390) | 0.2519 (0.02419) | 0.2715 (0.02404) | 0.0864 (0.02375)
  Week 1: number analyzed (Participants) | 80 | 78 | 80 | 78 | 82
  Week 1 | 0.1460 (0.03045) | 0.1890 (0.03065) | 0.1691 (0.03064) | 0.2039 (0.03074) | 0.0323 (0.03014)
  Week 2: number analyzed (Participants) | 78 | 74 | 76 | 78 | 80
  Week 2 | 0.1362 (0.03261) | 0.2010 (0.03302) | 0.1783 (0.03296) | 0.2104 (0.03279) | 0.0217 (0.03228)
  Week 3: number analyzed (Participants) | 76 | 71 | 75 | 78 | 78
  Week 3 | 0.1431 (0.03318) | 0.1860 (0.03372) | 0.1798 (0.03346) | 0.1739 (0.03321) | 0.0252 (0.03281)
  Week 4: number analyzed (Participants) | 73 | 70 | 75 | 76 | 79
  Week 4 | 0.1350 (0.03606) | 0.1928 (0.03654) | 0.1623 (0.03610) | 0.2134 (0.03594) | 0.0382 (0.03533)

13. Secondary Outcome: LS Mean Change From Baseline FVC to Average AUC0-12h FVC on Day 1 and at Week 4
Description: Forced spirometry maneuvers including the FVC were used to assess pulmonary function. Baseline FVC was defined as the value of FVC assessed 30 minutes before first administration and average AUC0-12h FVC was defined as area under the curve over 12 hours of the FVC, divided by 12 hours. Spirometry assessments were performed in accordance with ATS/ERS guidelines.
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | RPL554 0.375 mg | RPL554 0.75 mg | RPL554 1.5 mg | RPL554 3.0 mg | Placebo
Number analyzed (Participants) | 83 | 83 | 81 | 82 | 84
liters
  Day 1 | 0.0838 (0.02543) | 0.1294 (0.02543) | 0.1187 (0.02574) | 0.1514 (0.02558) | 0.0344 (0.02527)
  Week 4: number analyzed (Participants) | 74 | 71 | 76 | 78 | 78
  Week 4 | 0.0152 (0.03486) | 0.0838 (0.03529) | 0.0438 (0.03478) | 0.0982 (0.03443) | -0.0030 (0.03425)

14. Secondary Outcome: LS Mean Change From Baseline FVC to Morning Trough FVC at Weeks 1 to 4
Description: Forced spirometry maneuvers including the FVC were used to assess pulmonary function. Baseline FVC was defined as the value of FVC assessed 30 minutes before first administration and morning trough FVC was defined as the last pre-dose value. Spirometry assessments were performed in accordance with ATS/ERS guidelines.
Time Frame: Baseline (30 minutes before first administration on Day 1) and morning pre-dose on Weeks 1, 2, 3 and 4
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | RPL554 0.375 mg | RPL554 0.75 mg | RPL554 1.5 mg | RPL554 3.0 mg | Placebo
Number analyzed (Participants) | 83 | 83 | 81 | 82 | 84
liters
  Week 1: number analyzed (Participants) | 81 | 80 | 80 | 78 | 82
  Week 1 | -0.0159 (0.03028) | -0.0650 (0.03053) | -0.0887 (0.03053) | -0.0624 (0.03092) | -0.0617 (0.03008)
  Week 2: number analyzed (Participants) | 80 | 75 | 78 | 78 | 81
  Week 2 | -0.0647 (0.03190) | -0.0744 (0.03275) | -0.0458 (0.03231) | -0.0045 (0.03245) | -0.0614 (0.03170)
  Week 3: number analyzed (Participants) | 78 | 72 | 75 | 78 | 80
  Week 3 | -0.0966 (0.03354) | -0.0936 (0.03456) | -0.0857 (0.03410) | -0.0690 (0.03383) | -0.0969 (0.03318)
  Week 4: number analyzed (Participants) | 75 | 71 | 75 | 76 | 79
  Week 4 | -0.0390 (0.03323) | -0.0347 (0.03408) | -0.0570 (0.03344) | -0.0217 (0.03336) | -0.0198 (0.03264)

15. Secondary Outcome: Steady-State Plasma Concentrations of Tiotropium on Day 1 and at Week 2
Description: Blood samples were taken to determine steady-state plasma concentrations of tiotropium prior to and following 14 days of treatment with RPL554.
Time Frame: Pre-dose on Day 1 and Week 2
Population: The Pharmacokinetic (PK) analysis set included all randomized patients who had blood sampling performed and quantitative values of study treatment concentrations determined. Patients were classified according to actual treatment received for PK analysis set. One patient who was randomized to RPL554 0.375 mg group was dispensed wrong treatment kit and received RPL554 3 mg. Number of patients with values available at the specific visit were analyzed.
Measure: Mean (Standard Deviation); unit: picogram per milliliter (pg/mL)
Arm/Group | RPL554 0.375 mg | RPL554 0.75 mg | RPL554 1.5 mg | RPL554 3.0 mg | Placebo
Number analyzed (Participants) | 82 | 82 | 81 | 83 | 84
picogram per milliliter (pg/mL)
  Day 1: number analyzed (Participants) | 80 | 80 | 79 | 80 | 78
  Day 1 | 2.8 (1.18) | 2.1 (2.98) | 1.9 (1.4) | 2.4 (3.56) | 2.4 (3.06)
  Week 2: number analyzed (Participants) | 74 | 69 | 71 | 78 | 74
  Week 2 | 2.2 (3.85) | 2.3 (3.56) | 1.9 (1.58) | 2.0 (2.22) | 2.2 (2.13)

16. Secondary Outcome: Steady-State Plasma Concentrations of RPL554 at Week 2
Description: Blood samples were taken to determine steady-state plasma concentrations of RPL554 following 14 days of treatment with RPL554.
Time Frame: Pre-dose at Week 2
Population: The PK analysis set included all randomized patients who had blood sampling performed and quantitative values of study treatment concentrations determined. Patients were classified according to actual treatment received for PK analysis set. Number of patients with values available at the specific visit were analyzed.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | RPL554 0.375 mg | RPL554 0.75 mg | RPL554 1.5 mg | RPL554 3.0 mg | Placebo
Number analyzed (Participants) | 59 | 57 | 63 | 70 | 80
pg/mL | 37.3 (58.84) | 53.7 (51.71) | 107.9 (92.98) | 170.6 (154.3) | NA (NA)

17. Secondary Outcome: Number of Patients With Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was defined as any undesirable experience occurring to a patient, or worsening in a patient, whether considered related to the study medication or not. All AEs which started after the first dose of study treatment or started prior to first dose of study treatment and worsened, based on the Investigator's assessment of severity, on or after first dose of study treatment were considered to be treatment-emergent. A serious adverse event is any adverse experience that: results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; or other important medical events.
Time Frame: TEAEs were collected from the first dose of study treatment up to 1 week after the final study visit at Week 4, approximately 5 weeks.
Population: The safety analysis set included all randomized patients who received at least 1 dose of study treatment. One patient who was randomized to RPL554 0.375 mg group was dispensed wrong treatment kit and received RPL554 3 mg. Patients were classified according to actual treatment received for safety analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | RPL554 0.375 mg | RPL554 0.75 mg | RPL554 1.5 mg | RPL554 3.0 mg | Placebo
Number analyzed (Participants) | 82 | 83 | 81 | 83 | 84
Participants
  Any TEAE | 12 | 15 | 14 | 18 | 17
  Any TEAE leading to drug discontinuation | 2 | 3 | 0 | 0 | 1
  Any drug-related TEAE | 1 | 3 | 2 | 2 | 4
  Any serious TEAE | 0 | 1 | 0 | 2 | 0
  Any serious drug-related TEAE | 0 | 0 | 0 | 0 | 0
  Any serious TEAE leading drug discontinuation | 0 | 1 | 0 | 0 | 0
  Any TEAE leading to death | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: TEAEs were collected from the first dose of study treatment up to 1 week after the final study visit at Week 4, approximately 5 weeks.
Description: The safety analysis set included all randomized patients who received at least 1 dose of study treatment. One patient who was randomized to RPL554 0.375 mg group was dispensed wrong treatment kit and received RPL554 3 mg. Patients were classified according to actual treatment received for safety analysis set.
Groups:
- RPL554 0.375 mg: Patients were administered 0.375 mg RPL554 by jet nebulizer twice daily (morning and evening) for 4 weeks. Open-label tiotropium was administered once daily in the morning. Patients were classified according to actual treatment received for safety analysis set.
- RPL554 0.75 mg: Patients were administered 0.75 mg RPL554 by jet nebulizer twice daily (morning and evening) for 4 weeks. Open-label tiotropium was administered once daily in the morning. Patients were classified according to actual treatment received for safety analysis set.
- RPL554 1.5 mg: Patients were administered 1.5 mg RPL554 by jet nebulizer twice daily (morning and evening) for 4 weeks. Open-label tiotropium was administered once daily in the morning. Patients were classified according to actual treatment received for safety analysis set.
- RPL554 3.0 mg: Patients were administered 3.0 mg RPL554 by jet nebulizer twice daily (morning and evening) for 4 weeks. Open-label tiotropium was administered once daily in the morning. Patients were classified according to actual treatment received for safety analysis set.
- Placebo: Patients were administered placebo (matching with RPL554) by jet nebulizer twice daily (morning and evening) for 4 weeks. Open-label tiotropium was administered once daily in the morning. Patients were classified according to actual treatment received for safety analysis set.
Arm/Group | RPL554 0.375 mg | RPL554 0.75 mg | RPL554 1.5 mg | RPL554 3.0 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/82 | 0/83 | 0/81 | 0/83 | 0/84
Serious Adverse Events (participants affected / at risk) | 0/82 | 1/83 | 0/81 | 2/83 | 0/84
Other Adverse Events (participants affected / at risk) | 6/82 | 9/83 | 4/81 | 8/83 | 5/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RPL554 0.375 mg (N=82) | RPL554 0.75 mg (N=83) | RPL554 1.5 mg (N=81) | RPL554 3.0 mg (N=83) | Placebo (N=84)
Jaw fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alcohol abuse (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RPL554 0.375 mg (N=82) | RPL554 0.75 mg (N=83) | RPL554 1.5 mg (N=81) | RPL554 3.0 mg (N=83) | Placebo (N=84)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 0 (0) | 3 (3) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
One patient who was randomized to RPL554 0.375 mg group was dispensed wrong treatment kit and received RPL554 3 mg. Patients were classified according to randomized treatment for the FAS and actual treatment received for safety and PK analysis sets.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-12-05): https://cdn.clinicaltrials.gov/large-docs/79/NCT03937479/SAP_000.pdf
  • Study Protocol (2019-07-22): https://cdn.clinicaltrials.gov/large-docs/79/NCT03937479/Prot_001.pdf